CLINICAL TRIAL: NCT07322614
Title: Post-Market Clinical Trial of Neurorehabilitation With Mindlenses in Stroke Patients
Brief Title: Neurorehabilitation With Mindlenses in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RNT-CT#2
Record Dates: First submitted 2025-12-11; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: Post-Stroke Cognitive Rehabilitation, Prism Adaptation, Serious Games, MindLenses, Neurorehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: MindLenses Cognitive Rehabilitation (Experimental): Participants in the experimental arm receive cognitive rehabilitation using the MindLenses device, a medical device that integrates prism adaptation with serious game-based cognitive training. Each session begins with a prism-adaptation phase, during which participants perform visuomotor tasks under an optically induced visual deviation to promote sensorimotor recalibration. Following this phase, participants complete a series of adaptive serious games designed to stimulate cognitive domains commonly affected after stroke, including attention, visuospatial abilities, processing speed, and executive functions. The games progressively adjust their difficulty based on user performance, ensuring individualized cognitive stimulation. Training sessions are delivered under the supervision of rehabilitation professionals following a standardized protocol, with frequency and duration aligned with the rehabilitation center's clinical practice.
  Interventions: Device: MindLenses Cognitive Training
- Control: Standard Cognitive Rehabilitation (No Intervention): Participants in the control arm receive the standard cognitive rehabilitation program routinely provided in the clinical setting. This intervention consists of therapist-guided cognitive exercises targeting domains commonly affected after stroke, including attention, visuospatial abilities, processing speed, and executive functions. Sessions follow the center's established rehabilitation protocols and may include paper-and-pencil tasks, computerized cognitive exercises, visuospatial scanning activities, and structured problem-solving tasks. Training is administered by qualified rehabilitation professionals, with session frequency and duration consistent with usual clinical practice. No prism adaptation or gamified digital tasks are included in this arm.

INTERVENTIONS:
Device: MindLenses Cognitive Training — Cognitive rehabilitation delivered through the MindLenses medical device, which integrates prism adaptation with serious game-based cognitive exercises. Each session includes a visuomotor recalibration phase followed by adaptive game tasks targeting attention, visuospatial abilities, and executive functioning. Supervised by trained rehabilitation professionals according to a standardized protocol.
  Other Names: Prism Adaptation + Serious Games
  Arms: Experimental: MindLenses Cognitive Rehabilitation

SUMMARY:
This study aims to describe the use of MindLenses, a rehabilitation device that integrates prism adaptation with serious game-based cognitive exercises, in individuals undergoing cognitive rehabilitation after stroke. The intervention consists of structured sessions combining visuomotor recalibration and gamified cognitive tasks designed to target domains such as attention, visuospatial processing, and executive functions. The study examines changes in cognitive performance across the intervention period and documents the characteristics of the training program. The objective is to provide a detailed description of the implementation of MindLenses in a clinical rehabilitation setting and to characterize the cognitive domains addressed through the combined prism-adaptation and game-based approach.

DETAILED DESCRIPTION:
This clinical investigation aims to evaluate the safety and effectiveness of the MindLenses system, a medical device integrating prism adaptation with serious game-based cognitive training for post-stroke rehabilitation. The study includes two groups: an experimental group receiving the MindLenses intervention and a control group receiving standard cognitive and motor rehabilitation. The investigation focuses on device safety, changes in cognitive and motor performance, and measures related to usability and procedural feasibility.

Intervention Description:

The MindLenses intervention consists of a structured treatment session combining a prism-adaptation phase with adaptive serious games. During prism adaptation, participants perform visuomotor tasks under optically deviated vision to promote sensorimotor recalibration. The subsequent serious game phase provides exercises targeting attention, visuospatial abilities, executive functions, memory, and processing speed, with automatic difficulty adjustment based on performance. Sessions are delivered under therapist supervision and follow a standardized protocol.

Participants in the control group undergo standard clinical cognitive and motor rehabilitation, including paper-and-pencil tasks, visuospatial scanning, problem-solving activities, and conventional motor therapy. No prism-adaptation or serious-game elements are used in the control arm.

Assessments and Follow-Up:

All participants complete a comprehensive neuropsychological battery assessing memory, attention, language, executive functions, praxis and constructional abilities, intelligence, and visuospatial and visuoperceptual functions. Motor performance is evaluated using the Ashworth Scale (spasticity) and the Motor Assessment Scale (daily motor function).

Assessments are conducted at four time points:

Baseline (pre-treatment)

End of treatment

3-month follow-up

6-month follow-up

This schedule allows evaluation of both short-term outcomes and medium-term durability of rehabilitation effects.

Primary Endpoints:

The primary safety endpoint is the incidence of individual adverse events and device-related adverse events. Individual adverse events are recorded during treatment sessions, between sessions, and throughout the full follow-up period. Device-related events are recorded during sessions. The safety criterion is satisfied if both event rates remain within the acceptable thresholds defined in the device risk documentation.

The primary effectiveness endpoint is the change in cognitive and motor performance at the end of treatment. Cognitive indicators include standardized paper-and-pencil tests and additional clinical assessments; motor indicators include the Ashworth Scale and Motor Assessment Scale. The endpoint is met if improvements in the experimental group are not inferior to improvements observed in the control group.

Secondary Endpoints (Simplified):

Secondary endpoints provide additional evaluation of safety, usability, and operational feasibility of MindLenses. These include:

Technical success rate during session planning, execution, and reporting.

Procedural success rate at rehabilitation completion.

Occurrence of critical and non-critical procedural errors.

Occurrence of application errors reported by clinical staff.

Usability and logistical indicators (operator time, total therapy time, patient logistics).

Patient quality of life assessed via standardized questionnaire.

Significance:

This study provides a structured evaluation of a multimodal digital rehabilitation system integrating prism adaptation and serious games. By documenting safety, cognitive and motor outcomes, usability parameters, and clinical workflow integration, the investigation supports the validation of MindLenses as a medical device for post-stroke cognitive rehabilitation and contributes to the development of evidence-based digital neurorehabilitation strategies.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

* First ischemic or hemorrhagic stroke, with a minimum interval of 30 days from the acute event
* Presence of cognitive deficits identified during the pre-treatment neuropsychological assessment
* Ability to understand and sign informed consent and willingness to participate in follow-up assessments
* Age ≥ 18 years

Exclusion Criteria:

* Upper limb motor impairments preventing the use of a tablet
* Severe visual deficits affecting stimulus perception
* Concurrent neurological or psychiatric disorders
* Substance abuse
* Diagnosis of dementia
* Severe Wernicke's aphasia
* Age > 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Global Cognitive Function Change Over Time | Baseline, immediately after completion of treatment, 3-month follow-up, and 6-month follow-up
  Primary outcomes are changes in performance across a neuropsychological battery at baseline, post-treatment, 3- and 6-month follow-up. Measures include: Oxford Cognitive Screen (0-30), Raven's CPM (0-36), Digit Span (0-8), Corsi Block-Tapping (0-8), Rey 15-Word Test immediate (0-75) and delayed (0-15), Rey-Osterrieth Figure (0-36), Matrici Attentive (accuracy), Stroop interference (lower=better), Line Bisection deviation (lower=better), Bells Test (0-35), BADA Naming (accuracy), Phonemic and Semantic Fluency (correct words/60s), Copy of Drawings with (0-70) and without programming elements (0-12), VOSP (subtest scores), Buccofacial Apraxia Test (performance score). Higher scores indicate better performance unless noted.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Fondazione Santa Lucia, Roma, RM, Italy